CLINICAL TRIAL: NCT04880707
Title: Myogenous Face Pain Following Third Molar Extractions Under Intravenous Sedation
Brief Title: Twin Block, Pain Medications and Third Molar Extractions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Health Foundation (Other)
Responsible Party: Principal Investigator, Gayathri Subramanian, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro2020002007
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Acute Pain
Keywords: Twin block; Prescription opioids; Acute post-extraction pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Triple blind, randomized prospective pilot study comparing post wisdom molar extraction pain comparing placebo or Twin block local anesthetic nerve block injection
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, Twin block administrator and assessor assessing jaw muscle pain will all be unaware of whether the patient received sterile saline (placebo) or local anesthetic in the Twin Block injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Twin Block with Local Anesthetic (Active Comparator): Following lower third molar extraction under intravenous sedation, the patient randomized to this arm with receive the Twin block local anesthetic nerve block using the standard dental local anesthetic, i.e,. 2% lidocaine with 1:100,000 epinephrine, on the day after extraction, if the patient has pain greater than or equal to 5 on 10 in their jaw-closer muscles (Numerical Pain rating scale).
  Interventions: Drug: Twin block local anesthetic nerve block using standard dental anesthetic
- Twin Block with sterile normal saline (Placebo Comparator): Following lower third molar extraction under intravenous sedation, the patient randomized to this arm with receive the Twin block using sterile normal saline, on the day after extraction, if the patient has pain greater than or equal to 5 on 10 in their jaw-closer muscles (Numerical Pain rating scale).
  Interventions: Other: Twin block with placebo

INTERVENTIONS:
Drug: Twin block local anesthetic nerve block using standard dental anesthetic — 2% lidocaine with 1:100,000 epinephrine is the standard dental local anesthetic in universal use. This drug will be administered as the Twin block local anesthetic nerve block targeting the branches of the mandibular nerve supplying the temporalis and masseter muscles.
  Arms: Twin Block with Local Anesthetic
Other: Twin block with placebo — Instead of the standard dental anesthetic, sterile normal saline will be delivered using the Twin block injection
  Arms: Twin Block with sterile normal saline

SUMMARY:
Each year, over 3.5 million, mostly, healthy young adults, have their third molar teeth ('wisdom teeth') removed under sedation and are often given opioid prescriptions for managing their pain. Wisdom molar removal is one of the most common reasons for opioid prescriptions to be given to adolescents. There is a national thrust to reduce both the dose and the duration of such opioid prescriptions because even short-term opioid exposures increase risk for narcotic addiction and misuse. Non-opioid options to manage pain will still allow for sufficient pain control without risking addiction, and hence, a fundamental component of our response to combat the current national opioid crisis.

The investigators are going to study a promising option- the Twin Block dental anesthetic injection. The Twin block involves injecting the standard dental numbing medication in a way that 'numbs' the 'jaw-clencher' muscles on the side of the face. The investigators found that the Twin block relieved jaw pain stemming from these muscles, in a quick and sustained manner, even in patients whose pain following wisdom tooth removal primarily came from 'taut' and tender jaw-clencher muscles. However, what is not known is- how often do patients who have their wisdom teeth removed under sedation, end up in significant pain from taut and tender jaw-clencher muscles? Will using the twin block effectively reduce pain in such patients? In this pilot study, the investigators will examine wisdom molar extraction patients one day after their procedure. Those with significant pain (pain rated ≥ 5 on a 0-10 scale) in their jaw-clencher muscles, will get either the Twin block injection or a placebo. The investigators will track both 1) pain before and after the injection, and 2) pain medication usage over a 7-day period to see if both pain and opioid dosage come down with the Twin block. This study can support a simple, safe and inexpensive means to reduce pain after a common procedure.

DETAILED DESCRIPTION:
Annually, over 3.5 million predominantly young and healthy individuals undergo outpatient third molar tooth extractions and routinely receive postoperative opioid prescription (Moore, Nahouraii et al. 2006). This procedure is among the most prevalent instances of opioid prescriptions to adolescents and is the subject of a national debate, given the CDC's mandate for minimizing the number and duration of opioid prescriptions (Volkow, McLellan et al. 2011, Dowell, Haegerich et al. 2016, Moore, Dionne et al. 2016). Targeting such a prevalent practice by supplementing postoperative analgesia with non-opioid options as well as optimizing and tracking opioid usage will significantly reduce prescription opioid use/misuse. The Twin Block is a local anesthetic nerve block that eases muscle pain emanating from the jaw muscles and has been anecdotally shown to be effective in relieving post-operative pain in patients who developed muscle pain following third molar extractions. However, the incidence of acute muscle pain following third molar extractions is not well established. Accordingly, the aims of this study are two-fold:

A. Objectives This study has 2 objectives: 1) To estimate the incidence of acute muscle pain involving the temporalis and masseter muscles (the jaw closer muscles that are commonly implicated in resulting in jaw muscle pain), following third molar extractions and 2) Conduct a double-blind prospective study to compare the efficacy of Twin Block in relieving postextraction pain in those patients determined to experience muscle pain following the procedure B. Hypotheses / Research Question(s) Hypothesis 1: The incidence of post-third molar extraction muscle pain is at least 40% Hypothesis 2: Twin block reduces post-extraction muscle pain by 50% 1.2 Research Significance The twin block is a simple and effective local anesthetic nerve block for 'numbing' the innervation to the masseter and temporalis muscles, two key jaw clencher muscles, with emerging data corroborating efficacy in the diagnosis and management of both acute and chronic myogenous orofacial pain (Quek, Young et al. 2014, Ananthan et al. 2017). 1.3 Research Design and Methods The study is designed as a prospective evaluation of patients undergoing third molar extractions under intravenous sedation to identify those developing post-extraction muscle pain on the day following the procedure. Subsequently, such patients will be prospectively randomized to receive the Twin block to deliver either the dental local anesthetic or saline as a placebo. Post-injection muscle pain will be evaluated 15 minutes following the administration of the injection. All patients will be provided similar directions and prescriptions for pain management. All patients will be contacted to document/report their daily pain medications and queried one week after the extraction/s for their overall pain experience and any adverse effects from the injection.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring extraction/s of at least 1 lower wisdom (third) molar that is partially/fully 'impacted', under intravenous sedation, are eligible to participate in this study so long as they

  1. are older than 18 years of age,
  2. are healthy,
  3. have no cognitive/intellectual disability,
  4. have no past/recent pain or reduced range of motion in their jaw joint/ muscle complex, no trauma or surgery in their jaw region.
  5. have an electronic device such as a smart phone or a tablet/ computer with internet connection.
  6. are willing to participate in the study and not be excluded by the following criteria below.

Exclusion Criteria:

* Any patients, even if satisfying the criteria above, may not take part if they have any of the following:

  1. Compromised ability to guard their self-interest, for e.g., prisoners, children, pregnant women, patients with intellectual/cognitive disability are not enrolled in the study.
  2. Those patients who present with infection/inflammation involving the third molars slated for extractions, on the day of their procedure, may not take part in the study.
  3. In addition, those who have had opioid pain medication/s in the past to address short-term or long-standing pain, or those who are on long term prescription of anti-inflammatory pain medication, are unable to participate.
  4. Those with long standing pain of the jaw joint or muscles.
  5. Finally, those patients who are allergic to/unable to tolerate either the dental local anesthetic or its components, opioids, acetaminophen ('Tylenol') or ibuprofen ('Motrin' or 'Advil') also may not take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As reported by participant
Enrollment: 48 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Post-injection muscle pain | 15 minutes
  NRS pain scores before and 15 min after Twin block administration on day after procedure
Mean NRS pain score | one week
  Means NRS pain score by Day, comparing placebo and Twin block groups
Total prescription opioid consumption | one week
  Comparison of total prescription opioid consumption (mg) between placebo and Twin block groups

SECONDARY OUTCOMES:
Passive mouth opening | 15 min
  Comparison of passive mouth opening before and 15 min after Twin block administration on day after procedure
Passive mouth opening | one week
  Comparison of baseline and end-of-study passive mouth opening between Twin block and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri Subramanian, PhD, DMD, Principal Investigator — Rutgers School of Dental Medicine, Newark NJ
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
After anonymizing, IPD will be shared after the study is completed.
Supporting Information: Study Protocol
Time Frame: After study completion, upon review of request
Access Criteria: A written request will be evaluated and responded to.

REFERENCES:
- [Background] Quek S, Young A, Subramanian G. The twin block: a simple technique to block both the masseteric and the anterior deep temporal nerves with one anesthetic injection. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Sep;118(3):e65-7. doi: 10.1016/j.oooo.2014.01.227. Epub 2014 Feb 6. PMID 24703404
- [Result] Quek SYP, Gomes-Zagury J, Subramanian G. Twin Block in Myogenous Orofacial Pain: Applied Anatomy, Technique Update, and Safety. Anesth Prog. 2020 Jun 1;67(2):103-106. doi: 10.2344/anpr-67-01-03. PMID 32633773
- [Result] Kanti V, Ananthan S, Subramanian G, Quek SYP. Efficacy of the twin block, a peripheral nerve block for the management of chronic masticatory myofascial pain: A case series. Quintessence Int. 2017 Oct 6:725-729. doi: 10.3290/j.qi.a39094. Online ahead of print. PMID 28990015